CLINICAL TRIAL: NCT00423449
Title: A Phase I Clinical Trial of Vorinostat in Combination With Gemcitabine Plus Platinum in Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: Clinical Trial of MK0683 in Combination With FDA Approved Cancer Drugs in Patients With Advanced NSCLC (MK0683-058)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0683-058; 2006_528
Record Dates: First submitted 2007-01-17; First posted 2007-01-18 (Estimated); Results first posted 2011-08-02 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Advanced Stage IIIB/IV Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Vorinostat; Gemcitabine

ARMS (1):
- Vorinostat + Gemcitabine + Platinum-based agent (Experimental)
  Interventions: Drug: vorinostat; Drug: Gemcitabine; Drug: Platinum-based agent

INTERVENTIONS:
Drug: vorinostat — Dose escalation study: vorinostat 300-500 mg capsules once daily for 7-14 days in continuous cycles of 21 days
Drug: Gemcitabine — Dose escalation study: Gemcitabine 1000-1250 mg/m2 will be given for 2 days in each 21 day cycle
Drug: Platinum-based agent — Cisplatin IV 75 mg/m2 will be given for 1 day in each 21 day cycle or carboplatin dosed according to renal function.

SUMMARY:
This is a clinical trial to determine the safety and tolerability of MK0683 in combination with gemcitabine and cisplatin and/or carboplatin.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have a histologically-confirmed metastatic or locally advanced non-small cell lung cancer that has not been previously treated with systemic chemotherapy or has received non-platinum and non-gemcitabine based neoadjuvant or adjuvant chemotherapy if the last dose was at least 6 months prior to study enrollment

Exclusion Criteria:

* Patient who has had chemotherapy, radiotherapy, or biological therapy prior to entering the study, except for adjuvant or neoadjuvant chemotherapy, as allowed for treatment of a tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2007-03; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Groups:
- Vorinostat 300 7/21+ Gemcitabine 1000 + Cisplatin: Vorinostat 300 mg given the first 7 days of the 21 day cycle. Gemcitabine 1000 mg/m^2 given on days 3 & 10 of the 21 day cycle. Cisplatin 75 mg/m^2 given on day 3 of th 21 day cycle.
- Vorinostat 300 7/21+ Gemcitabine 1250 + Cisplatin: Vorinostat 300 mg given the first 7 days of the 21 day cycle. Gemcitabine 1250 mg/m^2 given on days 3 & 10 of the 21 day cycle. Cisplatin 75 mg/m^2 given on day 3 of th 21 day cycle.
- Vorinostat 400 7/21+ Gemcitabine 1250 + Cisplatin: Vorinostat 400 mg given the first 7 days of the 21 day cycle. Gemcitabine 1250 mg/m^2 given on days 3 & 10 of the 21 day cycle. Cisplatin 75 mg/m^2 given on day 3 of th 21 day cycle.
- Vorinostat 400 10/21+ Gemcitabine 1250 + Cisplatin: Vorinostat 400 mg given the first 10 days of the 21 day cycle. Gemcitabine 1250 mg/m^2 given on days 3 & 10 of the 21 day cycle. Cisplatin 75 mg/m^2 given on day 3 of th 21 day cycle.
- Vorinostat 400 14/21+ Gemcitabine 1250 + Cisplatin: Vorinostat 400 mg given the first 14 days of the 21 day cycle. Gemcitabine 1250 mg/m^2 given on days 3 & 10 of the 21 day cycle. Cisplatin 75 mg/m^2 given on day 3 of th 21 day cycle.
Period: Overall Study
Arm/Group | Vorinostat 300 7/21+ Gemcitabine 1000 + Cisplatin | Vorinostat 300 7/21+ Gemcitabine 1250 + Cisplatin | Vorinostat 400 7/21+ Gemcitabine 1250 + Cisplatin | Vorinostat 400 10/21+ Gemcitabine 1250 + Cisplatin | Vorinostat 400 14/21+ Gemcitabine 1250 + Cisplatin
Started | 4 | 6 | 17 | 27 | 7
Completed | 1 | 2 | 2 | 5 | 0
Not Completed | 3 | 4 | 15 | 22 | 7
Not completed — Clinical Adverse Event | 1 | 0 | 1 | 8 | 2
Not completed — Death | 1 | 0 | 2 | 1 | 1
Not completed — Progressive Disease | 1 | 3 | 8 | 11 | 4
Not completed — Laboratory Adverse Event | 0 | 1 | 2 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Vorinostat + Gemcitabine + Cisplatin
Arm/Group | All Participants
Number analyzed (Participants) | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.7 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 44

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-limiting Toxicities (DLT) Due to Vorinostat Administered in Combination With Standard Dose of Gemcitabine Plus Either Cisplatin or Carboplatin
Description: DLT = any Common Terminology Criteria for Adverse Events Grade 3/4 drug related non-hematologic toxicity EXCEPT Grade 3 nausea/vomiting responsive to therapy, Grade 3 Fatigue responsive to management, transient electrolyte disorders that were corrected, any Grade 4 drug related hematologic toxicity EXCEPT lymphopenia/neutropenia, unless the neutropenia was febrile and/or was an infection requiring treatment, OR Any Grade 4 neutropenia lasting >=7 days, failure of absolute neutrophil count or platelets to recover, or any drug-related AE that led to a dose reduction of >=1 study drugs.
Time Frame: every 21 days (every cycle), up to 126 days (6 cycles)
Measure: Number; unit: Participants
Arm/Group | Vorinostat 300 7/21+ Gemcitabine 1000 + Cisplatin | Vorinostat 300 7/21+ Gemcitabine 1250 + Cisplatin | Vorinostat 400 7/21+ Gemcitabine 1250 + Cisplatin | Vorinostat 400 10/21+ Gemcitabine 1250 + Cisplatin | Vorinostat 400 14/21+ Gemcitabine 1250 + Cisplatin
Number analyzed (Participants) | 4 | 6 | 17 | 27 | 7
Participants | 0 | 1 | 0 | 0 | 1

2. Secondary Outcome: Number of Participants With Clinical Adverse Experiences (Safety and Tolerability)
Description: An adverse experience (AE) was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the sponsor's product, whether or not considered related to the use of the product. Any worsening (any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which was temporally associated with the use of the sponsor's product, was also an adverse experience.
  The AEs could have been any grade from 1 to 5 in severity (mild, moderate, severe, life-threatening, death, respectively).
Time Frame: every 21 days (every cycle), up to 126 days (6 cycles)
Measure: Number; unit: Participants
Arm/Group | Vorinostat 300 7/21+ Gemcitabine 1000 + Cisplatin | Vorinostat 300 7/21+ Gemcitabine 1250 + Cisplatin | Vorinostat 400 7/21+ Gemcitabine 1250 + Cisplatin | Vorinostat 400 10/21+ Gemcitabine 1250 + Cisplatin | Vorinostat 400 14/21+ Gemcitabine 1250 + Cisplatin
Number analyzed (Participants) | 4 | 6 | 17 | 27 | 7
Participants | 4 | 6 | 17 | 27 | 7

3. Secondary Outcome: Number of Participants With Laboratory Adverse Experiences (Safety and Tolerability)
Description: An adverse experience was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the sponsor's product, whether or not considered related to the use of the product. Any worsening (any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which was temporally associated with the use of the sponsor's product, was also an adverse experience.
  The AEs could have been any grade from 1 to 5 in severity (mild, moderate, severe, life-threatening, death, respectively).
Time Frame: every 21 days (every cycle), up to 126 days (6 cycles)
Measure: Number; unit: Participants
Arm/Group | Vorinostat 300 7/21+ Gemcitabine 1000 + Cisplatin | Vorinostat 300 7/21+ Gemcitabine 1250 + Cisplatin | Vorinostat 400 7/21+ Gemcitabine 1250 + Cisplatin | Vorinostat 400 10/21+ Gemcitabine 1250 + Cisplatin | Vorinostat 400 14/21+ Gemcitabine 1250 + Cisplatin
Number analyzed (Participants) | 4 | 6 | 17 | 27 | 7
Participants | 2 | 4 | 7 | 13 | 2

4. Primary Outcome: Maximum Tolerated Dose of Vorinostat Administered in Combination With Standard Doses of Gemcitabine Plus Either Cisplatin or Carboplatin in Patients With Advanced Stage Non-Small Cell Lung Cancer Who Have Not Received Chemotherapy for Advanced Disease
Description: Maximum tolerated dose (MTD) was defined as the highest dose level in which fewer than 2 patients among the first 6 enrolled experience a DLT (as defined in Outcome Measure 1) during the first cycle of treatment.
  The MTD was 400 mg for up to 10 days in 21-day cycles.
Time Frame: every 21 days (every cycle), up to 126 days (6 cycles)
Measure: Number; unit: mg
Arm/Group | All Participants
Number analyzed (Participants) | 61
mg | 400

ADVERSE EVENTS:
Arm/Group | MK-0683 300 mg x 7d/21d + Gemcitabine 1000 mg/m^2 + Cisplatin | MK-0683 300 mg 7d/21d + Gemcitabine 1250 mg/m^2 + Cisplatin | MK-0683 400 mg 7d/21d + Gemcitabine 1250 mg/m^2 + Cisplatin | MK-0683 400 mg 10d/21d + Gemcitabine 1250 mg/m^2 + Cisplatin | MK-0683 400 mg 14d/21d + Gemcitabine 1250 mg/m^2 + Cisplatin
Serious Adverse Events (participants affected / at risk) | 3/4 | 4/6 | 10/18 | 18/27 | 4/7
Other Adverse Events (participants affected / at risk) | 4/4 | 6/6 | 17/18 | 27/27 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-0683 300 mg x 7d/21d + Gemcitabine 1000 mg/m^2 + Cisplatin (N=4) | MK-0683 300 mg 7d/21d + Gemcitabine 1250 mg/m^2 + Cisplatin (N=6) | MK-0683 400 mg 7d/21d + Gemcitabine 1250 mg/m^2 + Cisplatin (N=18) | MK-0683 400 mg 10d/21d + Gemcitabine 1250 mg/m^2 + Cisplatin (N=27) | MK-0683 400 mg 14d/21d + Gemcitabine 1250 mg/m^2 + Cisplatin (N=7)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (3) | 0 (0) | 0 (0) | 4 (5) | 2 (5)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Device occlusion (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Disease progression (General disorders) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
Hyperthermia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Bronchopneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood potassium increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bladder dilatation (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (3) | 1 (1) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-0683 300 mg x 7d/21d + Gemcitabine 1000 mg/m^2 + Cisplatin (N=4) | MK-0683 300 mg 7d/21d + Gemcitabine 1250 mg/m^2 + Cisplatin (N=6) | MK-0683 400 mg 7d/21d + Gemcitabine 1250 mg/m^2 + Cisplatin (N=18) | MK-0683 400 mg 10d/21d + Gemcitabine 1250 mg/m^2 + Cisplatin (N=27) | MK-0683 400 mg 14d/21d + Gemcitabine 1250 mg/m^2 + Cisplatin (N=7)
Anaemia (Blood and lymphatic system disorders) | 4 (11) | 6 (14) | 11 (33) | 23 (72) | 4 (27)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (4) | 2 (4) | 6 (22) | 9 (43) | 4 (21)
Lymphopenia (Blood and lymphatic system disorders) | 2 (2) | 2 (10) | 1 (1) | 8 (34) | 4 (13)
Neutropenia (Blood and lymphatic system disorders) | 2 (7) | 4 (10) | 12 (51) | 15 (69) | 5 (20)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (7) | 6 (15) | 10 (29) | 18 (55) | 5 (29)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 5 (15) | 0 (0)
Bundle branch block right (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Coronary artery insufficiency (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ototoxicity (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (5) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (1) | 4 (4) | 1 (1)
Aerophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aphthous stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (4) | 2 (2) | 8 (12) | 9 (11) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 4 (5) | 10 (11) | 3 (6)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 5 (12) | 11 (21) | 19 (43) | 4 (15)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 4 (6) | 7 (12) | 13 (33) | 5 (9)
Asthenia (General disorders) | 4 (8) | 6 (10) | 12 (21) | 22 (39) | 5 (18)
Chest pain (General disorders) | 1 (3) | 1 (1) | 3 (4) | 4 (4) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Generalised oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperthermia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 3 (4) | 2 (2) | 2 (2) | 6 (8) | 1 (1)
Cytolytic hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (3) | 3 (3) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pseudomonal bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (6) | 1 (2) | 3 (6) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 1 (3) | 1 (1) | 4 (9) | 3 (6)
Blood bicarbonate decreased (Investigations) | 1 (1) | 2 (8) | 0 (0) | 2 (10) | 2 (4)
Blood creatinine increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 3 (5) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Blood magnesium increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Blood potassium increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 2 (3) | 0 (0)
Blood sodium decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 0 (0)
Blood urea decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Carbon dioxide decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Creatinine renal clearance decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram PR prolongation (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (2) | 2 (7) | 3 (9) | 7 (27) | 3 (5)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 3 (3) | 1 (2)
Lymphocyte count decreased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 2 (2) | 5 (13) | 6 (15) | 1 (6)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 5 (11) | 10 (20) | 2 (5)
Protein total decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Protein urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 3 (3) | 0 (0) | 7 (8) | 2 (6)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 2 (3) | 2 (3) | 8 (10) | 16 (22) | 5 (9)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyperalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercreatininaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (5) | 2 (14) | 3 (9) | 9 (34) | 3 (7)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (3) | 1 (1) | 7 (22) | 3 (7)
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 (3) | 2 (2) | 0 (0) | 7 (16) | 2 (5)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (4) | 0 (0) | 6 (16) | 2 (8)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (6) | 0 (0) | 7 (20) | 2 (7)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 0 (0) | 5 (5) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (4) | 1 (2) | 4 (10) | 3 (6)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 2 (9) | 2 (5) | 8 (16) | 3 (7)
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 3 (3) | 2 (2) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (2)
Formication (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 1 (3)
Motor dysfunction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (5) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 4 (4) | 2 (2) | 2 (2)
Confusional state (Psychiatric disorders) | 1 (3) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3) | 4 (4) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 3 (4) | 2 (2) | 2 (3)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 4 (6) | 5 (5) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (8) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 6 (6) | 7 (13) | 3 (3)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 0 (0)
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subcutaneous nodule (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Extremity necrosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Peripheral coldness (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication guidelines.